CLINICAL TRIAL: NCT04067323
Title: Study on the Efficacy of MCT (Medium-chain Triglycerides) Oil Consumption on Nutritional Status and Blood Lipid Profile in Overweight and Obese (Class II) Vietnamese Women
Brief Title: Improvement of Nutritional Status and Blood Lipid Profile by Using MCT Oil on Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition, Vietnam (Other Government)
Responsible Party: Principal Investigator, Tu Nguyen Song, Head of Division Planning, National Institute of Nutrition, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nortalic-NIN 176
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Obesity Adult Onset; Lipid Metabolism Disorder
Keywords: obesity; medium chain triglycerides; blood lipid profile
MeSH Terms: conditions — Lipid Metabolism Disorders; Obesity | interventions — Soybean Oil

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, community-controlled intervention trial. A screening survey will be used to recruit women aged from 20 to 45 considered overweight and obese within a city of Bac Giang province, Viet Nam, during which subjects will conduct nutritional status and determine whether overweight or obesity and eligible criteria. Subjects then will be randomly allocated to receive 1 of 2 treatment sequences, with a balanced number of subjects assigned to each dietary treatment (either MCT oil or Soya bean oil/soy oil mixed in yogurt together with their standard meals (lunch) daily) over a period of 4 months and their blood lipid and nutritional profiles checked.
Who Masked: Participant, Investigator
Masking Description: The list of participants will be randomly coded and divided two group will be sealed. This envelop will stored by the head of National Institute of Nutrition, Vietnam. The investigators will be not known who the participants consume test product or placebo product during the recruiting stage and whole intervention period. The oil product will be packed in the same bottles (only different from coloring the label bottles), manufactured by Nortalic, Vietnam.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCT consumption (Placebo Comparator): 20g soy oil (containing mainly long chain triglycerides - LCT) together with 100g yogurt) will be provided in lunch-daily meal for a period of 4 months.
  Interventions: Dietary Supplement: Soya bean oil
- MCT consumption (Experimental): 20g MCT oil (containing 100% MCT) together with 100g yogurt) will be provided in lunch-daily meal for a period of 4 months.
  Interventions: Dietary Supplement: MCT oil

INTERVENTIONS:
Dietary Supplement: Soya bean oil — Participants will consume soya bean oil together with yogurt in lunch daily meals and be monitored side effects and diarrhea. Then they will be evaluated anthropometric index, body compositions and blood lipid profile after 2 months (T1) and 4 months (T2) intervention. This product is composed of 12% total energy intake of participants.
  Arms: LCT consumption
Dietary Supplement: MCT oil — Participants will consume MCT oil together with yogurt in lunch daily meals and be monitored side effects and diarrhea. Then they will be evaluated anthropometric index, body compositions and blood lipid profile after 2 months (T1) and 4 months (T2) intervention. This product is composed of 12% total energy intake of participants.
  Arms: MCT consumption

SUMMARY:
The purpose of this study is to examine whether MCT oil is effective in the change of blood lipid profile and body compositions on overweight or obese women aged 20-45.

DETAILED DESCRIPTION:
A randomized, double-blinded, community-controlled trial will be conducted to verify the effects of MCT oil on blood lipid profile and body compositions. 160 overweight or obese female subjects aged 20-45 years with body weight index [25 kg/m2 ≤ body mass index (BMI) < 40 kg/m2] will be recruited. The subjects will visit the research site for 4 times. On the first visit, the participants will be recruited to determine exact BMI, age range and eligible criteria. On the second visit, the recruited participants will be randomly assigned to consume a test or placebo product [test product: plain yogurt blending MCT oil; placebo product: plain yogurt blending soy oil (mainly long chain triglycerides - LCT)] and ingest the assigned product in daily lunch meals for 4 months. On the next 3 visits (at baseline, 2 months and 4 months after intervention), the 12-hr fasting blood samples test will be conducted to check lipid blood profile and glucose; the body compositions and anthropometric index will be measured.

Plans for site monitoring will be conducted by the independent supervisors from the National Institute of Nutrition's Experts who come from the different departments of NINVietnam and the experts of the collaborator for each visiting day and on the days when the participants receive products (every 10 days). In the site research, multiply supervised and cross-over staff will be implemented (staff from NINVietnam, Center of Disease Control branch, Medical Center of Province and Local Ward Health Stations). For following the consumed products, each participant will daily self-note in a designed notebook (trained before delivering products). If there is any different information between the staff and others, information will be checked again. The participants, consuming at least 90% the total amount of product, will be considered as complete intervention and will be analyzed.

Data will be collected by questionnaire and checked again in the same day of collecting. Investigators will request and correct at the site research if any suspicious answer or missing data. The Body composition analyzer SC-330 TANITA scale will be checked and corrected before using. Each 100 subjects, this scale will be checked and corrected again. Data are reported as mean ± standard deviation, compared between 2 arms and in each group between baseline time and 2 or 4 months interventions.

ELIGIBILITY:
Inclusion Criteria:

In Recruiting investigation:

* Citizen women from 20 to 45 years old in the selected area
* Subjects at risk of being overweight, obese or having BMI > 23 (self-estimate)
* Voluntarily agree to participate

In Intervention study:

* Eligible criteria from screening investigation
* Body Mass Index from 25.0 to 39.99 kg/m2
* Voluntarily agree to participate

Exclusion Criteria:

In Recruiting investigation:

* History/presence of high blood pressure or diabetes
* Pregnant or breastfeeding women

In Intervention study:

* Medication known to affect body weight
* Chronic diseases
* Plan to move out of the area within next 6 months
* Plan to have pregnancy within next 4-5 months

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women, in Vietnam, who are in reproductive age usually following the intervention more than men and they are also more interested in their appearance. Investigators hope the participants will complete this study with at least withdrawal numbers.
Enrollment: 161 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Blood lipid profile, i.e. changes of blood lipid measurements | over 2 and 4 months intervention
  Blood samples are drawn after 12 hours and not over 16 hours overnight fasting and at least 24 hours of alcohol abstinence and collected in Heparin-containing (BD Vacutainer USA) tubes. Blood samples will consist of Cholesterol, Triglyceride, HDL-cholesterol and LDL-cholesterol and evaluated by The National Cholesterol Education Program (NCEP), e.g. JAMA, 2001. 285(19): p. 2486-2497

SECONDARY OUTCOMES:
Body Mass Index, i.e. changes of Body Mass Index (BMI) | over 2 and 4 months
  Weight is measured in kg with one decimal value by the Body composition analyzer SC-330 TANITA scale. Height is measured by wooden stadiometer with exactly 0.1cm. Then, these raw data will be calculated to BMI (kg/m^2). All data will be measured at the time T0 (at baseline), T1 (after 2 months) and T2 (after 4 months).
Waist - Hip Ratio, i.e. changes of Waist - Hip Ratio (WHR) | over 2 and 4 months
  Waist and hip circumferences are measured in cm, with one decimal value are by tape. Participants wear light clothes while measuring.
Percentage of total fat, i.e. changes of percentage of total fat | over 2 and 4 months
  Measurement of total fat percentage is measured by the Body composition analyzer SC-330 TANITA scale.
Fat mass, i.e. changes of fat mass | over 2 and 4 months
  Measurement of fat mass is measured in kg, with one decimal by the Body composition analyzer SC-330 TANITA scale.

OTHER OUTCOMES:
Fasting blood glucose, i.e. changes of fasting blood glucose | at baseline time, over 2 and 4 months
  Blood samples were drawn after 12 hours and not over 16 hours overnight fasting and at least 24 hours of alcohol abstinence and collected in Heparin-containing tubes and analyzed at the same time with blood lipid profile. Fasting blood glucose will be measured by Beckman Coulter AU 680 automated analyzer and evaluated by American Diabetes Association: e.g. Diabetes Care, 2010: p. 33 (suppl): S11-S69.

CONTACTS AND LOCATIONS:
Overall Officials: Tu S Nguyen, PhD., Principal Investigator — National Institute of Nutrition, Vietnam
Locations (1):
- National Institute of Nutrition, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] St-Onge MP, Bosarge A, Goree LL, Darnell B. Medium chain triglyceride oil consumption as part of a weight loss diet does not lead to an adverse metabolic profile when compared to olive oil. J Am Coll Nutr. 2008 Oct;27(5):547-52. doi: 10.1080/07315724.2008.10719737. PMID 18845704
- See also: Click here for more information about the organisation in which this study is conducted. The Division of Planning is responsible to plan and implement the project — http://viendinhduong.vn/en/home.html